CLINICAL TRIAL: NCT05662748
Title: Use of the Closure Device in Patient With Percutaneous Transfemoral Aortic Valve Replacement
Brief Title: Comparison Between Manta and Prostar Closure Devices
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jörg Schröder, PD Dr. med Jörg Schröder, RWTH Aachen University
Other Study IDs: RWTH AachenU
Record Dates: First submitted 2022-11-15; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Aortic Valve Stenosis
Keywords: Closure
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pro Star: patient received Pro Star Device
  Interventions: Device: Transfemoral aortic valve replacement
- MANTA: Patient received MANTA Device
  Interventions: Device: Transfemoral aortic valve replacement

INTERVENTIONS:
Device: Transfemoral aortic valve replacement — aortic valve replacement

SUMMARY:
Use of the closure device in patient with percutaneous transfemoral aortic valve replacement

DETAILED DESCRIPTION:
The advent of endovascular, transcatheter aortic valve replacement (TAVR), and mechanical circulatory support has offered new, minimally invasive therapeutic options that are rapidly becoming standard of care. These percutaneous transfemoral interventions require large-bore catheters and have created challenges for femoral arterial access management. Current approaches include surgical cut-down with arterial puncture under direct vision, and suture-based "pre-closure." Surgical cut-down is associated with longer procedural time, increased patient discomfort, deeper anesthesia, risk of wound complications including infection, and slower ambulation. The pre-closure technique overcomes many of the disadvantages of surgical cut-down but can be technically demanding, time consuming, and associated with a significant failure rate. Recent randomized TAVR trials have reported major vascular complications in 6% to 8% . Furthermore, a study on the 2 suture-based closure techniques for management of TAVR access reported a 20% vascular complication rate despite being used by experienced operators . Currently, the majority of access site complications result from failed arteriotomy closure . The percutaneous MANTA Vascular Closure Device (VCD) (Essential Medical Inc., Malvern, Pennsylvania) is a novel collagen-based technology dedicated to closure of largebore arteriotomies . The MANTA VCD underwent prospective multicenter evaluation for Conformitä Europäenne (CE) mark approval in the first detailed report of outcomes achieved with a dedicated large-bore vascular closure device Contrary to the aforementioned TAVR procedures, mechanical circulatory support therapy can be extended up to several days on the intensive care ward. Data on such delayed closure with is lacking. This registry is therefore aimed to document the initial experiences of delayed closure of a femoral large bore access with vascular closure devices in patients with an TAVR device.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for treatment with the TAVR device 2. Decision to use the Manta or the Prostar closure device on a clinical base by the treating physician 3. Signed informed consent

Exclusion Criteria:

* Male or female aged < 18 2. Pregnant and lactating females 3. Patient has been committed to an institution by legal or regulatory order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with planned treatment of aortic valve replacement will be asked to participate in the observational study
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Safety endpoints during index hospitalisation | 2018 - 2020
  Major vascular complications,
Safety endpoints during index hospitalisation ( bleeding) | 2018-2020
  life-threatining-, major bleeding
Safety endpoints during index hospitalisation ( death ) | 2018-2020
  death

SECONDARY OUTCOMES:
efficacy endpoints during index hospitalisation - (hemotasis) | 2018-2020
  hemotasis in angiogram
efficacy endpoints during index hospitalisation ( device failure) | 2018-2020
  device failure
efficacy endpoints during index hospitalisation ( bail-out ) | 2018-2020
  need for stent-graft

OTHER OUTCOMES:
preperation time | 2018-2020
  preperation time for closure

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Schröder, Principal Investigator — Universitätsklinikum Aachen Medizinische Klinik 1; Michael Lehrke, Principal Investigator — Universitätsklinikum Aachen Medizinische Klinik 1
Locations (1):
- Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Study results will be published in an appropriate scientific journal. The Ethics Committee will be informed about the study results.